CLINICAL TRIAL: NCT06297421
Title: Efficacy and Safety of Fecal Microbiota Transplantation for the Treatment of Irritable Bowel Syndrome With Diarrhea (IBS-D) and Mental Health Comorbidity in Young Adults: A Randomized, Double-blind, Placebo Controlled Study
Brief Title: Efficacy and Safety of FMT for the Treatment of IBS-D and Mental Health Comorbidity in Young Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Chen Ye, M.D., Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SZYY20240229IBS-D
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Irritable Bowel Syndrome With Diarrhea; Fecal Microbiota Transplantation; Mental Health Issue
Keywords: Irritable Bowel Syndrome with Diarrhea; Fecal Microbiota Transplantation; Randomized Controlled Study; Mental Health Comorbidity; Young Adults
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (Experimental): Oral Fecal Microbiota Transplantation Capsule Take 40 capsules daily, 20 capsules in the morning and 20 capsules in the evening for 3 consecutive days. This is a cycle. Take it for three consecutive cycles.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Placebo (Placebo Comparator): Oral Placebo Capsule Take 40 capsules daily, 20 capsules in the morning and 20 capsules in the evening for 3 consecutive days. This is a cycle. Take it for three consecutive cycles.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Oral Fecal Microbiota Transplantation Capsule
  Arms: Fecal Microbiota Transplantation
Procedure: Placebo — Oral Placebo Capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Fecal Microbiota Transplantation compared with placebo in the treatment of Irritable Bowel Syndrome With Diarrhea (IBS-D) and Mental Health Comorbidity in Young Adults.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent, be able to comply with the protocol and be able to carry out related procedures, including the completion of diary during the induction period and throughout the study period.
2. Age between 18 and 29 years old (including two-end values, based on the date of signing the Master Informed consent), regardless of gender.
3. IBS-D patients with clinical symptoms meeting the Rome IV definition, that is, the course of disease for at least 6 months, repeated abdominal pain in the past 3 months, an average of at least 1 day per week, combined with two or more of the following conditions: (a) Abdominal pain is related to defecation; （b） Abdominal pain accompanied by changes in the frequency of defecation; （c） Abdominal pain accompanied by changes in fecal trait. When abnormal stool occurred in the last 3 months, the proportion of abnormal stool was >25% for Bristol fecal trait type 6 or 7, and <25% for Bristol fecal trait type 1 or 2；and a Hamilton Depression Scale score: 20-34 and/or a Hamilton Anxiety Scale score: 14-28 were evaluated as depressed or anxious patients;
4. Colonoscopy has been completed within 12 months before the run-in period. The ileocecal part should be observed during endoscopy, and the ileocecal flap image recording should be included in the report. They may be included if one of the following conditions is met: (i) The colonoscopy report is normal; (ii) Abnormalities reported by colonoscopy, such as hemorrhoids and intestinal polyps (diameter ≤5mm and number ≤3), were determined by the investigator to be eligible for inclusion; (iii) Colonoscopy reported that the diameter of intestinal polyps was >5mm or the number of intestinal polyps was >3; after endoscopic treatment, the diameter of residual intestinal polyps was ≤5mm and the number of intestinal polyps was ≤3, and the investigators determined that they could be included in the group.
5. The patient had not used any relief drugs or analgesics in the 14 days prior to randomization.
6. During the period from the signing of the master informed consent to the end of the final study visit, patients agreed to maintain their usual diet and lifestyle, such as no changes in dietary structure or exercise patterns.

Exclusion Criteria:

1. Patients with constipated, mixed and amorphous IBS.
2. Patients with organic gastrointestinal diseases were excluded from the following conditions: superficial gastritis, grade I erosive gastritis, chronic atrophic gastritis found by endoscopy but judged by the investigator to be eligible for admission (for example, no mucosal erosion or bleeding under endoscopy, and no abdominal distension, epigastric pain, acid reflux and other symptoms).
3. Parenteral diseases of the digestive system such as tuberculous peritonitis, pancreatitis, cirrhosis, and biliary tract diseases are present, except for fatty liver disease that has not progressed to hepatitis, and gallstones that lack related symptoms.
4. Known to have lactose intolerance and celiac disease.
5. There are other systemic diseases, including serious diseases of the heart, lungs and kidneys, malignant tumors, autoimmune diseases, metabolic diseases (such as diabetes, diseases affecting thyroid function), reproductive system diseases (such as ovarian cysts, endometriosis, severe dysmenorrhea requiring medical treatment), etc.
6. Previous history of abdominal and pelvic surgery, except appendectomy, caesarean section but no intestinal complications, hernia repair.
7. Patients with severe mental disorders other than depression and anxiety.
8. Fecal examination results showed occult blood (+) and above (except for cases caused by hemorrhoids or female menstrual periods) or white blood cells (+) and above, and were judged by the investigator to be clinically significant.
9. People who are positive for antibodies against hepatitis C virus (HCV), or human immunodeficiency virus (HIV), or syphilis, or hepatitis B surface antigen (HBsAg) and need antiviral therapy at the screening stage.
10. Laboratory tests showed significant abnormalities, and the investigator determined that the patient's participation in the study may compromise his or her safety, including but not limited to: (i) Creatinine ≥1.5 times the upper limit of normal (ULN); (ii) AST≥2 times upper limit of normal (ULN) and/or ALT≥2 times upper limit of normal (ULN) and/or total bilirubin ≥1.5 times upper limit of normal (ULN).
11. A history of drug or alcohol abuse.
12. Even with the help of liquids, patients are unable to take oral solid dosage forms.
13. Allergic to experimental drugs, rescue drugs and their ingredients.
14. During the trial, drugs that affect gastrointestinal movement and function cannot be discontinued, It includes antibiotics (such as erythromycin), drugs that regulate intestinal microecology (such as bifidobacterium), parasympathetic inhibitors (such as scopolamine, atropine, belladona, etc.), muscle relaxants (such as succinylcholine), antidiarrheal agents (such as loperamide, montmorillonite powder, etc.), opioids, drugs that inhibit gastric acid secretion, etc.
15. A woman who is pregnant or breastfeeding.
16. At the time of the trial, both the patient and his partner were unable or unwilling to use reliable contraception to prevent pregnancy, or the female or male patient's partner had a recent pregnancy plan.
17. Have participated in any clinical trial and used the experimental drug or device within 3 months prior to signing the informed consent.
18. The patient had previously participated in a clinical study of FMT and received FMT therapy.
19. According to the judgment of the investigator, the participants are not suitable to participate in this clinical trial.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients Who Were Composite Weekly Responders | 1-12 weeks
  A patient is categorized as a composite weekly responder if the patient achieved the prespecified response displayed in the following for at least 50% of the weeks during the interval from weeks 1-12.
  Abdominal pain response: a decrease in the weekly average of worst abdominal pain (as measured by the 11-point NRS-scale) in the past 24 hours score of at least 30% compared with baseline.
  Stool consistency response: a 50% or greater reduction in the number of days per week with at least one stool that has a consistency of Type 6 or 7 (as measured by the Bristol Stool Form Scale) compared with baseline.
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v5.0 | 1-52weeks
  The number of participants with adverse events both severe and non-severe, assessed for severity based on the 5-grade criteria set by the NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
Percentage of Patients Who Were Composite Weekly Responders | 1-8weeks、1-4weeks、5-8weeks、9-12weeks
  A patient is categorized as a composite weekly responder if the patient achieved the prespecified response displayed in the following for at least 50% of the weeks during the interval from weeks 1-8、weeks 1-4、weeks 5-8 or weeks 9-12.
  Abdominal pain response: a decrease in the weekly average of worst abdominal pain (as measured by the 11-point NRS-scale) in the past 24 hours score of at least 30% compared with baseline.
  Stool consistency response: a 50% or greater reduction in the number of days per week with at least one stool that has a consistency of Type 6 or 7 (as measured by the Bristol Stool Form Scale) compared with baseline.
Percentage of Patients Who Were Abdominal Pain Weekly Responder | 1-12weeks、1-8weeks、1-4weeks、5-8weeks、9-12weeks
  A patient is categorized as an abdominal pain weekly responder if the patient achieved prespecified response, i.e. a decrease in the weekly average of worst abdominal pain (as measured by the 11-point NRS-scale) in the past 24 hours score of at least 30% compared with baseline on at least 50% of weeks during the interval from weeks 1-12、weeks 1-8、weeks 1-4、weeks 5-8 or weeks 9-12.
Percentage of Patients Who Were Stool Consistency Weekly Responder | 1-12weeks、1-8weeks、1-4weeks、5-8weeks、9-12weeks
  A patient is categorized as an stool consistency weekly responder if the patient achieved prespecified response, i.e. a 50% or greater reduction in the number of days per week with at least one stool that has a consistency of Type 6 or 7 (as measured by the Bristol Stool Form Scale) compared with baseline on at least 50% of weeks during the interval from weeks 1-12、weeks 1-8、weeks 1-4、weeks 5-8 or weeks 9-12.
Percentage of Patients Who Were Abdominal Bloating Weekly Responder | 1-12weeks、1-8weeks、1-4weeks、5-8weeks、9-12weeks
  A patient is categorized as an abdominal bloating weekly responder if the patient achieved prespecified response, i.e. a decrease in the weekly average of worst abdominal bloating (as measured by the 11-point NRS-scale) in the past 24 hours score of at least 30% compared with baseline on at least 50% of weeks during the interval from weeks 1-12、weeks 1-8、weeks 1-4、weeks 5-8 or weeks 9-12.
Percentage of Participants Who Were Responders in IBS Symptoms Relief Scale | 1-12weeks、1-8weeks、1-4weeks、5-8weeks、9-12weeks
  Relief of IBS symptoms was assessed once weekly by patients answering the IBS Symptoms Relief Scale in the electronic diary. Responders were defined as patients with a weekly response of "Yes" to relief of their IBS symptoms for at least 50% of weeks during the interval from weeks 1-12、weeks 1-8、weeks 1-4、weeks 5-8 or weeks 9-12.
Change from Baseline in the Weekly Average of Worst Abdominal Pain in the Past 24 hours | 1-12 weeks
  Symptoms of abdominal pain were measured by the 11-point NRS-scale, where 0 corresponded to no abdominal pain and 10 corresponded to worst imaginable abdominal pain. A negative change from Baseline indicates the abdominal pain decreased.
Change from Baseline in the Number of Days per Week with at Least One Stool with Consistency of Type 6 or 7 | 1-12 weeks
  Patients recorded the number of days per week with at least one stool with consistency of Type 6 or 7 during weeks 1-12. Stool consistency was measured by the Bristol Stool Form Scale.
Change from Baseline in the Number of Stools of Type 6 or 7 per Week | 1-12 weeks
  Patients recorded the number of stools of Type 6 or 7 every day during weeks 1-12. Stool consistency was measured by the Bristol Stool Form Scale.
Change from Baseline in the Weekly Average of Worst Abdominal Bloating in the Past 24 Hours Score | 1-12 weeks
  Symptoms of abdominal bloating were measured by the 11-point NRS-scale, where 0 corresponded to no abdominal bloating and 10 corresponded to worst imaginable abdominal bloating. A negative change from Baseline indicates the abdominal bloating decreased.
Change from baseline in Irritable Bowel Syndrome Severity Scale (IBS-SSS) Scores | week4、week8、week9、week12、week20、week28、week36、week44、week52
  The IBS Symptom Severity Score is produced from 5 symptom responses on the questionnaire, the total score with a possible range of scores from 0 to 500. A negative change from Baseline indicates that IBS symptom severity improved.
Change from baseline in Irritable Bowel Syndrome Quality of Life Scale (IBS-QoL) Total Scores | week4、week8、week9、week12、week20、week28、week36、week44、week52
  The IBS-QoL consists of 34 items each with a 5-point response scale, where 1 generally represents better responses on items and 5 represents worse responses. The individual responses to the answered items were summed and standardized for a total score and then transformed to a 0- to 100- point scale (0=worst; 100=better) for ease of interpretation. A positive change from Baseline indicates that quality of life improved.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong, China